CLINICAL TRIAL: NCT03823196
Title: Bioavailability, Pharmacokinetic and Mechanistic Study of Sinetrol® Xpur, a Polyphenol-rich Ingredient: an Open-label Study on Overweight Volunteers During a Chronical Supplementation and a Post-supplementation Follow-up
Brief Title: Bioavailability, Pharmacokinetic and Mechanistic Study of Sinetrol® Xpur, a Polyphenol-rich Ingredient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fytexia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SNTOL2019
Record Dates: First submitted 2019-01-23; First posted 2019-01-30 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum900 (Experimental): The arm will receive 900 mg of Sinetrol® Xpur, a blend of citrus and guarana extracts, daily for 16 weeks
  Interventions: Dietary Supplement: Verum900
- Verum1800 (Experimental): The arm will receive 1800 mg of Sinetrol® Xpur, a blend of citrus and guarana extracts, daily for 16 weeks
  Interventions: Dietary Supplement: Verum1800

INTERVENTIONS:
Dietary Supplement: Verum900 — Sinetrol® Xpur is a blend of polyphenol-rich extracts from grapefruit, guarana seed, sweet orange and blood orange. Daily dosage is 900 mg for 16 weeks
  Other Names: Sinetrol® Xpur
  Arms: Verum900
Dietary Supplement: Verum1800 — Sinetrol® Xpur is a blend of polyphenol-rich extracts from grapefruit, guarana seed, sweet orange and blood orange. Daily dosage is 1800 mg for 16 weeks
  Other Names: Sinetrol® Xpur
  Arms: Verum1800

SUMMARY:
The purpose of the study is to investigate the metabolization and the bioavailability of bioactive compounds from Sinetrol® Xpur, a polyphenol-rich ingredient, during a 16-week long chronical supplementation. It will be investigated the mechanism of action in adipocyte cells to try to explain the beneficial effects of the ingredient on body composition, especially on both abdominal subcutaneous and visceral fat mass.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male and female with 30% min. and 70% max. of each sex, aged range: 20-50 years old
4. Overweight BMI range (27-30)
5. Having a total fat mass (BIA assessment) ≥ 25% for men and ≥ 32% for women
6. In good general health as evidenced by medical history
7. Ability to take oral medication and be willing to adhere to the regimen
8. Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration

Exclusion Criteria:

1. Metabolic/Chronic disorders or any kind of disease
2. Current use of any medication or food supplement
3. Have in the past been in long-term antibiotherapy (1 month or more) and/or a regular antiobiotherapy in the past 12 months
4. Former obese with a history of yoyo-effect
5. Have been involved in a weight loss program in the past 12 months or subjected to a weight reduction surgery
6. Pregnancy or lactation, or women wanting to have a baby
7. Menopausal women
8. Known allergic reactions to components of the supplement, i.e., orange, grapefruit, guarana and/or caffeine
9. Having started or quit smoking
10. Having a high alcohol consumption

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Change in urine polyphenol metabolites excretion after acute and chronic ingestion of the ingredient | Week 1 and Week 16
Change in plasma polyphenol metabolites concentration after acute and chronic ingestion of the ingredient | Week 1 and Week 16

SECONDARY OUTCOMES:
Change in fecal microbiota composition | Week 1, Week 8, Week 16 and Week 20 (follow-up)
Change in blood microbiota composition | Week 1, Week 8, Week 16 and Week 20 (follow-up)
Change in adipose tissue microbiota composition | Week 1 and Week 16
Change in adipose tissue lipolysis assessed with glycerol concentration | Week 1 and Week 16
Change in adipose tissue lipolysis assessed with free fatty acids concentration | Week 1 and Week 16
Change in adipocytes diameters in adipose tissue | Week 1 and Week 16
Change in adipose tissue secretion profile assessed by leptin concentration | Week 1 and Week 16
Change in adipose tissue secretion profile assessed by adiponectin concentration | Week 1 and Week 16
Change in total fat mass assessed by DXA | Week 1, Week 16 and Week 20 (follow-up)
Change in total fat-free mass assessed by DXA | Week 1, Week 16 and Week 20 (follow-up)
Change in abdominal fat mass assessed by MRI | Week 1 and Week 16
Change in abdominal subcutaneous fat mass assessed by MRI | Week 1 and Week 16
Change in abdominal visceral fat mass assessed by MRI | Week 1 and Week 16
Change in energy expenditure assessed by indirect calorimetry | Week 1, Week 16 and Week 20 (follow-up)
Change in safety variables assessed by blood pressure variation (systole and diastole in mmHg) | Week 1 and Week 16
Change in safety variables assessed by heart rate variation | Week 1 and Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Pedro E Alcaraz Ramon, Principal Investigator — UCAM
Locations (1):
- UCAM, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muralidharan J, Romain C, Chung L, Alcaraz P, Martinez-Noguera FJ, Keophiphath M, Lelouvier B, Ancel P, Gaborit B, Cases J. Effect of Sinetrol(R) Xpur on metabolic health and adiposity by interactions with gut microbiota: a randomized, open label, dose-response clinical trial. Nutr Metab (Lond). 2024 Oct 16;21(1):83. doi: 10.1186/s12986-024-00851-7. PMID 39415279
- [Derived] Muralidharan J, Romain C, Bresciani L, Mena P, Angelino D, Del Rio D, Chung LH, Alcaraz PE, Cases J. Nutrikinetics and urinary excretion of phenolic compounds after a 16-week supplementation with a flavanone-rich ingredient. Food Funct. 2023 Nov 27;14(23):10506-10519. doi: 10.1039/d3fo02820h. PMID 37943075